CLINICAL TRIAL: NCT04711824
Title: Phase I/II Study of Stereotactic Radiosurgery With Concurrent Administration of DNA Damage Response (DDR) Inhibitor (OLAparib) Followed by Adjuvant Combination of DuRvalumab (MEDI4736) and Physician's Choice Systemic Therapy in Subjects With BreAst Cancer Brain Metastases
Brief Title: Study of Stereotactic Radiosurgery With Olaparib Followed by Durvalumab and Physician's Choice Systemic Therapy in Subjects With Breast Cancer Brain Metastases
Acronym: SOLARA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Colette Shen (Other)
Collaborators: AstraZeneca (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Colette Shen, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN BRE18-360
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Brain Metastases, Adult
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — olaparib; Radiosurgery; durvalumab; Paclitaxel; 130-nm albumin-bound paclitaxel; eribulin; Carboplatin; Cisplatin; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Treatment Arm (Experimental): Cycle 1 of study treatment will consist of Olaparib twice daily concurrently with stereotactic radiosurgery (SRS). Olaparib will start one week prior to SRS and continue during and following SRS (1-5 fractions) for up to 28 days total. Once the subject has recovered from SRS, Cycle 2 will be initiated with physician's choice systemic therapy and durvalumab. Cycle 2+ will equal 21 days. During Cycles 2 and 3, physician's choice systemic monotherapy will be given along with durvalumab. Each cycle will last 21 days. Imaging to evaluate intracranial and extracranial disease will be performed after Cycle 3, and subjects with response will continue with the systemic therapy and durvalumab until progression (intracranial or extracranial), unacceptable toxicity or death.
  Interventions: Drug: Olaparib; Radiation: Stereotactic Radiosurgery; Drug: Durvalumab; Drug: Physicians Choice systemic chemotherapy

INTERVENTIONS:
Drug: Olaparib — Olaparib 100-300 mg twice daily up to 28 days concurrently with stereotactic radiosurgery. Three dose levels of olaparib will be explored in the Phase I portion. Olaparib will start one week prior to SRS and continue during and following SRS for up to 28 days total. One cycle will be given.
  Other Names: Lynparza
Radiation: Stereotactic Radiosurgery — SRS 1-5 fractions will be given per institutional standards
  Other Names: SRS
Drug: Durvalumab — Durvalumab 1120 mg IV over 60 minutes Day 1 of each cycle 21 day cycle.
  Other Names: Imfinzi
Drug: Physicians Choice systemic chemotherapy — Olaparib: 300mg PO BID; Days 1-21 Paclitaxel: 80 mg/m2 IV over 60 min; Day 1 and 8 Nab-paclitaxel:100 mg/m2 IV over 30 min; Day 1 and 8 Eribulin: 1.4 mg/m2 IV over 2-5 min; Day 1 and 8 Carboplatin: AUC 2 mg/ml/min IV over 30-60 min; Day 1 and 8 Cisplatin: 75 mg/m2 IV over 30-60 min; Day 1 Capecitabine: 1000 mg/m2 PO BID; Days 1-14 Gemcitabine: 1000 mg/m2 IV over 30 min; Day 1 and 8 Gemcitabine + Carboplatin: 1000mg/m2 IV over 30-60 min; Day 1 and 8
  Other Names: Olaparib; Paclitaxel; Nab-paclitaxel; Eribulin; Carboplatin; Cisplatin; Capecitabine; Gemcitabine

SUMMARY:
This study is a Phase I/II study evaluating the safety and effectiveness of focused radiation therapy (radiosurgery) together with olaparib, followed by immunotherapy, for patients with brain metastases from triple negative or BRCA-mutated breast cancers.

This study will have a Phase I portion in which subjects will be enrolled based on 3+3 dose escalation rules. Three dose levels of olaparib will be studied.

Cycle 1 of study treatment will consist of Olaparib given twice daily concurrently with stereotactic radiosurgery (SRS). Olaparib will start one week prior to SRS and continue during and following SRS (1-5 fractions) for up to 28 days total. The number of doses of Olaparib will be dependent on how long it takes a subject to recover from SRS (ideally the subject will be off steroids, if they are required, at the start of Cycle 2, with exceptions outlined later in this section).

Once the subject has recovered from SRS (based on investigator discretion) that will be considered the DLT period. Cycle 2 will be initiated with physician's choice systemic therapy and durvalumab. Cycle 2+ will equal 21 days. During Cycles 2 and 3, physician's choice systemic monotherapy will be given along with durvalumab per protocol. Each cycle will last 21 days. Imaging to evaluate intracranial and extracranial disease will be performed after Cycle 3, and subjects with response will continue with the systemic therapy and durvalumab until progression (intracranial or extracranial), unacceptable toxicity or death.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Subject has histologically confirmed diagnosis of breast cancer per AJCC 8th edition meeting any of the following criteria: 1) triple negative, defined as ER/PR expression <10% and HER2-negative, with any BRCA status; or 2) HER2-negative (with ER/PR expression >=10% with germline or somatic BRCA mutation.
3. Subject has diagnosis of new brain metastasis by MRI, with a plan to undergo stereotactic radiosurgery (SRS) (up to 15 untreated metastases and at least 1 metastasis with maximum dimension > 5mm). Patients are permitted to have undergone recent craniotomy and resection of metastasis/metastases if at least 1 other intact metastasis or gross residual tumor planned for definitive SRS is present. Patients may have had prior SRS as long as the previously treated brain metastases are stable and not planned for additional therapy. Re-irradiation of a lesion previously treated with SRS is not allowed. Discrete dural lesions are allowed.
4. Subject may have other sites of extracranial metastatic disease (does not need to be stable, as long as no signs of impending visceral crisis).
5. Subjects may have had prior systemic therapy other than combination DDR inhibitor (PARP inhibitor) and immune checkpoint inhibitor (i.e., prior PARP inhibitor without concurrent immune checkpoint inhibitor, or prior immune checkpoint inhibitor without concurrent PARP inhibitor, are allowed).
6. Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within 28 days prior to registration.
7. Body weight >30 kg (for durvalumab monotherapy or durvalumab combination).
8. Subject has life expectancy > 16 weeks.
9. Age ≥ 18 years at the time of consent.
10. Prior systemic cancer treatment must be completed at least 7 days prior to treatment and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline.
11. Subject is willing and able to provide blood and tissue samples for correlative research activities, if applicable.
12. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined in the table below:

    * Platelets ≥100 x 109/L
    * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
    * Hemoglobin (Hgb) ≥ 10 g/dL with no blood transfusion in the past 28 days
    * Calculated creatinine clearance ≥ 51 mL/min
    * Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) ≤ 2.5 × ULN unless liver metastases are present in which case they must be ≤ 5x ULN
    * Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) Alanine aminotransferase (ALT) ≤ 2.5 × ULN unless liver metastases are present in which case, they must be ≤ 5x ULN
    * International Normalized Ratio (INR) or Prothrombin Time (PT)
    * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN; Patients taking warfarin may participate in this study; however, it is recommended that INR be monitored carefully at least once per week for the first month, then monthly if the INR is stable.
13. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1. Postmenopausal is defined as:

    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1-year interval since last menses
    * Surgical sterilisation (bilateral oophorectomy or hysterectomy)
14. Female patients of childbearing potential must be willing to abstain from heterosexual activity or to use 2 highly effective methods of contraception as described in the protocol from the time of informed consent until 3 months after treatment discontinuation.
15. Male patients must be willing to abstain from heterosexual activity or use a condom during treatment and for 3 months after treatment discontinuation. See the protocol for additional information.
16. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
17. Other inclusion criteria as specified by drug manufacturer for specific investigational drug(s), and/or required to specify disease status etc.

Exclusion Criteria:

1. Subject has evidence of diffuse symptomatic leptomeningeal carcinomatosis.
2. Subject has symptomatic brain metastases requiring immediate surgical resection within 1 week.
3. Subject has evidence of intracranial hemorrhage or signs of impending herniation.
4. Subject has had prior whole brain radiation therapy. Prior SRS to brain metastases is allowed as long as previously treated lesions are stable and not planned for further therapy.
5. Subject has had prior extracranial radiation therapy within 3 weeks of study initiation unless palliative.
6. Subject has signs of impending visceral crisis.
7. Subject has a history of severe brain injury.
8. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 7 days prior to the first dose of study drug. If sufficient wash-out time has not occurred (defined as 5 half-lives for the prior anti-cancer therapy), a longer wash-out period will be required, as agreed by sponsor-investigator and the site investigator. Concurrent use of hormonal therapy for non-cancer-related conditions is acceptable.
9. Subject with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
10. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
11. Subject has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
12. Subject has a history of interstitial lung disease.
13. Subject has a diagnosis of primary immunodeficiency.
14. Subject must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating study therapy.
15. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
16. Subject is pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
17. Subject is not eligible for sequential MRI or CT evaluations.
18. Subject with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
19. Subject unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
20. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
21. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
22. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
23. Participation in another clinical study with an investigational product during the last 4 weeks. NOTE: Subjects that consented to the sub-study may enroll in the primary therapeutic study if they meet all eligibility criteria outlined in Section 3.1.
24. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study. NOTE: Subjects that consented to the sub-study may enroll in the primary therapeutic study if they meet all eligibility criteria outlined in Section 3.1.
25. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

    * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor-investigator.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the sponsor-investigator.
26. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
27. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product (IP). NOTE: Resection of brain metastasis and local surgery of isolated lesions for palliative intent is acceptable.
28. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the sponsor-investigator
    * Patients with celiac disease controlled by diet alone
29. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
30. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    * Adequately treated carcinoma in situ without evidence of disease.
31. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
    * Steroids used to treat edema from SRS as per protocol.
32. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
33. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
34. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
35. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤ Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
36. Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

    * tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice),
    * hepatitis B (known positive HBV surface antigen (HBsAg) result),
    * hepatitis C, or
    * human immunodeficiency virus (positive HIV 1/2 antibodies).

NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for ≥ 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.

Eligibility Criteria for surgical sub-study

Inclusion Criteria

Subjects planned for surgical resection of their brain metastasis must meet the following criteria:

1. Subject is planned for surgical resection of their brain metastasis. NOTE: subjects with acutely symptomatic brain metastasis requiring surgical resection within 1 week are not eligible for the sub-study.
2. Subject meets inclusion criteria #1, 2, 4, 6, 8-16 above.1 Female patients of child-bearing potential and male patients must be willing to abstain from heterosexual intercourse or use contraception as described in protocol.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the surgical sub-study:

1. Subject has acutely symptomatic brain metastasis requiring surgical resection within 1 week.
2. Subject meets criteria #1, 2, 4, 7-17, 20-25, 27-28, 30, 33-34 above from section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | 4 weeks
  Phase I: frequency and severity of adverse events will be measured using common toxicity criteria for adverse events version 5.
Intracranial Disease control rate | 6 months
  Phase II: Intracranial disease control rate will be defined as the percentage of subjects with [complete response (CR) + partial response (PR) + stable disease] per RANO-BM criteria at 6 months after study treatment initiation.

SECONDARY OUTCOMES:
Intracranial disease progression free survival per RANO-BM | 2 years
  Intracranial progression free survival (PFS) is defined as time from the day of study treatment initiation until evidence of disease progression per RANO-BM or death from any cause.
Overall survival | 2 years
  Overall survival (OS) will be calculated starting from the day of study treatment initiation until death from any cause.
Intracranial response rate | 2 years
  Intracranial response rate will be measured by RANO-BM criteria.
Extracranial response rate per RECIST 1.1 | 2 years
  Extracranial response rate will be measured by RECIST 1.1 criteria.
Intracranial disease progression free survival per iRANO | 2 years
  Intracranial progression free survival (PFS) is defined as time from the day of study treatment initiation until evidence of disease progression per iRANO or death
Extracranial disease progression free survival per RECIST | 2 years
  Extracranial disease progression free survival (PFS) is defined as time from the day of study treatment initiation until evidence of disease progression per RECIST 1.1 or death
Extracranial disease progression free survival per iRECIST | 2 years
  Extracranial disease progression free survival (PFS) is defined as time from the day of study treatment initiation until evidence of disease progression per iRECIST or death
Extracranial response rate per iRECIST criteria. | 2 years
  Extracranial response rate will be measured by iRECIST criteria.
Intracranial response rate per iRANO criteria. | 2 years
  Intracranial response rate will be measured by iRANO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Colette Shen, M.D., Ph.D, Principal Investigator — University of North Carolina, Chapel Hill
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Memorial Healthcare System, Hollywood, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No